CLINICAL TRIAL: NCT05726266
Title: Effect and Safety of Listening to Music or Audiobooks as a Coadjunvant Treatment for Chronic Pain Patients Under Opioid Treatment: A Single-Center, Open-Label, Parallel Groups, Controlled, Randomized Pilot Clinical Trial
Brief Title: Effect and Safety of Listening to Music for Chronic Pain Relief
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sebastian Videla (Other)
Responsible Party: Sponsor-Investigator, Sebastian Videla, Head of the Clinical Research Support Unit, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UB-FCL-MUSIC 2022
Record Dates: First submitted 2023-01-25; First posted 2023-02-13 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain
Keywords: Music; Chronic Pain; Chronic Non-Cancer Pain
MeSH Terms: conditions — Chronic Pain | interventions — Music Therapy; Sound Recordings

STUDY DESIGN:
Intervention Model Description: All included patients must be under regular (maintenance) opioid treatment for at least one month before randomization. Included patients will be randomized (1:1) either to the control (audiobooks) or to the experimental (music) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group (Experimental): Patients randomized to this group will listen daily to a musical playlist for 30 - 60 minutes in a row through a mobile device. This will be performed in addition to the opioid treatment.
  Interventions: Other: Music
- Audiobooks Group (Placebo Comparator): Patients randomized to this group will listen to an audiobook daily for 30 - 60 minutes in a row through a mobile device. This will be performed in addition to the opioid treatment.
  Interventions: Other: Audiobook

INTERVENTIONS:
Other: Music — Patients will listen daily to a musical playlist for 30 - 60 minutes in a row; the psychologist will set up a music playlist according to the patient's individual interests. Patients will be asked to focus on this activity, that is, without performing any other activity simultaneously.
  Arms: Music Group
Other: Audiobook — Patients will listen daily to an audiobook for 30 - 60 minutes in a row; the psychologist will set up a list of audiobooks according to the patient's individual interests. Patients will be asked to focus on this activity, that is, without performing any other activity simultaneously.
  Arms: Audiobooks Group

SUMMARY:
Chronic pain is a multidimensional pathological condition that reduces patients' quality of life and interferes with their daily family and work activities.

Opioids are the most powerful analgesics in the treatment of pain. They are used as a basic analgesic treatment for managing patients with chronic pain and as an analgesic treatment for managing breakthrough pain.

Chronic administration of opioids can cause significant side effects (e.g., dependence, constipation) and tolerance to their analgesic effects, limiting their use. Different behavioral therapies (e.g., mindfulness and cognitive therapy) have been proposed to potentiate the analgesic effects of opioids and, consequently, reduce the dose and the appearance of adverse effects. One of the proposed approaches consists of listening to music therapeutically as a cognitive tool that modulates attention and regulates mood. Some studies provide evidence that music can reduce opioid requirements in patients with chronic pain. On the other hand, both opioids and music activate brain circuits for reward, reinforcement, and motivation.

Preliminary results obtained by our research group in animal models suggest that listening to music can reduce the appearance of a withdrawal syndrome after chronic administration of opioids.

Our working hypothesis is that multimodal therapy, based on listening to music as an adjuvant treatment to regular analgesic treatment with opioids, reduces pain intensity and its harmful effects in patients diagnosed with chronic non-cancer pain. Hence, the daily amount of opioids taken will be reduced, as well as the likelihood of developing opioid tolerance, dependence, and other opioid-related adverse events. At the same time, these patients' emotional well-being and quality of life will improve.

This is a parallel-group, open-label, single-center randomized, pilot, controlled clinical trial that aims to evaluate the effect and safety of music as a coadjuvant treatment for chronic non-cancer pain.

DETAILED DESCRIPTION:
Chronic non-cancer pain (CNCP) is defined as pain lasting from three to six months or persisting for longer than expected for tissue healing or underlying disease resolution [López, 2014]. Other authors define it as pain lasting for more than three months, continuously or intermittently, present more than five days a week, with moderate or high intensity on the visual analog scale (VAS), and/or impairing one's functional capacity [Guerra de Hoyos, 2014].

The World Health Organization (WHO) estimates that 20% of the world population suffers from chronic pain to some degree [Turk, 2011]. Moreover, CNCP impacts patients' quality of life substantially, affecting physical and psychosocial dimensions and interfering with daily-life activities. It also poses a heavy burden on health and social security services by increasing healthcare and economic aid demand for lost days at work [Breivik, 2013; Zimmer, 2021; Hopkins, 2022].

The main objective of the treatment is to maintain physical and mental functionality while improving quality of life. This may require a multimodal approach, including, in addition to medication, other interventions such as psychological therapy, active physiotherapy, movement therapy, or percutaneous electrostimulation, among others [Turk; 2011]. However, opioid use has been on the rise in the last few years, and its use is not free from adverse events.

Our working hypothesis is that a multimodal therapy, based on listening to music as a coadjuvant treatment to maintenance analgesic treatment with opioids, reduces pain intensity in patients diagnosed with CNCP. As a result, the daily amount of opioids taken will be reduced, as well as the likelihood of developing opioid tolerance, dependence, and other opioid-related adverse events. At the same time, these patients' emotional well-being and quality of life will improve.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≥18 years of age.
* Diagnosed with Chronic Non-Oncological Pain.
* Under regular (maintenance) opioid treatment for at least one month.
* Patients who sign the written informed consent.

Exclusion Criteria:

* Pregnant or lactating women.
* History of an organic brain disorder or substance abuse/dependence.
* History of Psychotic disorder, bipolar disorder, and/or intellectual disability.
* Patients at risk of opioid addiction.
* Patients that the Pain Clinic physician or psychologist believe will not comply with the study treatment/procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured by the Visual Analog Scale | 4 weeks
  The Visual Analog Scale is a continuous variable on a 10 cm line representing "no pain" (0 cm) to "worst imaginable pain" (10 cm).
  We will consider as responders those patients with a ≥30% reduction in the "maximum pain intensity in the last 24 hours" at any time during the study compared to the baseline score (study start visit) for at least 3 consecutive days.
Pain intensity differences from baseline during the 4 weeks of treatment | 4 weeks
  We will assess the mean pain intensity differences from baseline during the 4 weeks of treatment. These mean pain intensity differences will be used to obtain the sum of pain intensity differences (by calculating the area under the time-analgesic effect curve).
Scores on the McGill Multidimensional Pain Questionnaire | 4 weeks
  The McGill Multidimensional Pain Questionnaire scores range from 0 (No Pain) to 78 (Severe Pain). Changes between the baseline and end-of-treatment scores will be assessed.

SECONDARY OUTCOMES:
Change in pain intensity considering alternative definitions of responder (also measured by the Visual Analog Scale) | 4 weeks
  Other definitions of responder will be considered for capturing different response nuances:
  * Alternative Responder (AR) 1: ≥50% reduction in the "maximum pain intensity (MPI) in the last 24h" at any given time during the study compared to the baseline score for at least 3 consecutive days.
  * AR2: ≥30% reduction in the "current pain" at any given time during the study compared to the baseline score for at least 3 consecutive days.
  * AR3: ≥50% reduction in the "current pain" at any given time during the study compared to the baseline score for at least 3 consecutive days.
  * AR4: ≥30% reduction in the "MPI in the last 24h" AND in the "current pain" at any given time during the study compared to the baseline score for at least 3 consecutive days.
  * AR5: ≥50% reduction in the "MPI in the last 24h" AND in the "current pain" at any given time during the study compared to the baseline score for at least 3 consecutive days.
Requirement of rescue analgesia | 4 weeks
  As an alternative way of measuring pain intensity. Therefore, we will consider another definition of responder:
  • Alternative Responder 6: patients who do not require rescue analgesia.
Change of status according to the Hospital Anxiety and Depression Scale (HADS) scores between the baseline and end-of-treatment visits. | 4 weeks
  The Hospital Anxiety and Depression Scale (HADS) is composed of 2 subscales, one for depression and the other for anxiety. Each subscale consists of 7 items; each item score ranges from 0 (best result possible) to 3 (worst result possible). A final subscale score is achieved by summing the items scores.
  Scores in each subscale ranging from 0 to 7 denote normal levels of anxiety/depression; scores ranging from 8 - 10 denote borderline cases; scores ranging from 11 to 21 denote abnormal cases.
Mean Total Mood Disturbance (TMD) scores (measured by the Profile of Mood States [POMS]) between the baseline and end-of-treatment visits. | 4 weeks
  The Profile of Mood States (POMS) questionnaire assesses six mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. High vigor scores reflect a good mood or emotion, and low scores in the other subscales reflect a good mood or emotion. The total mood disturbance (TMD) score is computed by adding the five negative subscale scores (tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion) and subtracting the vigor score. Higher TMD scores indicate a greater degree of mood disturbance.
Mean change in the Patient Global Impression of Change (PGIC) scores between the baseline and end-of-treatment visits. | 4 weeks
  The Patient Global Impression of Change (PGIC) is a self-reported 7-point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Mean change in the Short-Form 36 (SF-36) scores between the baseline and end-of-treatment visits. | 4 weeks
  The Short-Form 36 (SF-36) consists of 36 questions meant to reflect 8 domains of health, including physical functioning, physical role, pain, general health, vitality, social function, emotional role, and mental health. Scores range from 0 (maximum disability) to 100 (no disability).
Change in the EuroQoL - 5 Dimensions - 5 Levels (EQ-5D-5L) scores between the baseline and end-of-treatment visits. | 4 weeks
  The EuroQoL - 5 Dimensions - 5 Levels (EQ-5D-5L) comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Number of adverse events by treatment arm. | 4 weeks
  Overall number of AEs in each group
Number of side effects derived from opioid use (UKU scale) | 4 weeks
  These will be assessed by the Udvalg für Kliniske Undersøgelser (UKU) Side Effect Rating Scale, a comprehensive rating scale that includes 48 individual side effects that can be grouped into the four main dimensions of psychic, neurological, autonomic and other side effects.
Number of adverse events related to the treatments under study (music therapy or audiobooks). | 4 weeks
  Number of adverse events considered as treatment-emergent adverse events.
Mean change in the Opioid Risk Tool (ORT) score | 4 weeks
  The Opioid Risk Tool (ORT) is a brief, self-report screening tool to assess the risk for opioid abuse among individuals prescribed opioids for treatment of chronic pain. Total scores of 3 or lower indicate low risk for future opioid abuse; 4 to 7 indicate moderate risk; and a score of 8 or higher indicate a high risk.
Mean change in the Revised Screener and Opioid Assessment for Patients with Pain (SOAPP-R) questionnaire score. | 4 weeks
  The Revised Screener and Opioid Assessment for Patients with Pain (SOAPP-R) is a 24-question questionnaire created to help determine how much monitoring a patient on long-term opioid therapy might require. Questions are scored form 0 (best result) to 4 (worst result). A total score of 18 or higher is considered positive.

CONTACTS AND LOCATIONS:
Overall Officials: Ancor S Alfonso, MD, Principal Investigator — Anesthesiologist at Bellvitge University Hospital
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The datasets used or analyzed during the study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Turk DC, Wilson HD, Cahana A. Treatment of chronic non-cancer pain. Lancet. 2011 Jun 25;377(9784):2226-35. doi: 10.1016/S0140-6736(11)60402-9. PMID 21704872
- [Background] Zimmer Z, Fraser K, Grol-Prokopczyk H, Zajacova A. A global study of pain prevalence across 52 countries: examining the role of country-level contextual factors. Pain. 2022 Sep 1;163(9):1740-1750. doi: 10.1097/j.pain.0000000000002557. Epub 2021 Dec 15. PMID 35027516
- [Background] Hopkins RE, Degenhardt L, Campbell G, Farnbach S, Gisev N. "Frustrated with the whole system": a qualitative framework analysis of the issues faced by people accessing health services for chronic pain. BMC Health Serv Res. 2022 Dec 31;22(1):1603. doi: 10.1186/s12913-022-08946-8. PMID 36587208
- [Background] Breivik H, Eisenberg E, O'Brien T; OPENMinds. The individual and societal burden of chronic pain in Europe: the case for strategic prioritisation and action to improve knowledge and availability of appropriate care. BMC Public Health. 2013 Dec 24;13:1229. doi: 10.1186/1471-2458-13-1229. PMID 24365383
- [Derived] Grau-Sanchez J, Serrano A, Villoria J, Carnaval T, Porto MF, Zapata L, Flores-Garcia M, Segura E, Garrido-Pedrosa J, Rodriguez-Fornells A, Fernandez-Duenas V, Videla S. Effect and safety of listening to music or audiobooks as a coadjuvant treatment for chronic pain patients under opioid treatment: a study protocol for an open-label, parallel-group, randomised, controlled, proof-of-concept clinical trial in a tertiary hospital in the Barcelona South Metropolitan area. BMJ Open. 2023 Sep 11;13(9):e074948. doi: 10.1136/bmjopen-2023-074948. PMID 37696633
- See also: Guerra de Hoyos, 2014 — https://www.juntadeandalucia.es/export/drupaljda/salud_5af1956f88676_dolor_cronico_julio_2014.pdf
- See also: López, 2014 — https://sanidad.castillalamancha.es/sites/sescam.castillalamancha.es/files/documentos/farmacia/dolor_cronico_0.pdf